CLINICAL TRIAL: NCT02566655
Title: Phase I Clinical Trial To Evaluate The Intravenous Infusion Of Autologous Fucosylated Bone Marrow Mesenchymal Cells Therapy In Patients With Established Osteoporosis and Low Impact Fractures
Brief Title: Clinical Trial of Intravenous Infusion of Fucosylated Bone Marrow Mesenchyme Cells in Patients With Osteoporosis
Acronym: CSM/OP/2011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other); Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other); Spanish National Health System (Other); Public Health Service, Murcia (Other); BIONAND, Universidad de Málaga, IBIMA, Ciber-bbn (Unknown); Grupo de Tecnología Sanitaria CIBER-BBN, Inst. Biomecánica de Valencia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/OP/2011; 2012-005814-20 (EudraCT Number)
Record Dates: First submitted 2015-01-30; First posted 2015-10-02 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2019-11

CONDITIONS: Osteoporosis; Spinal Fractures
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fucosylated MSC for Osteoporosis (Experimental): Autologous Bone Marrow fucosylated mesenchymal stem cells will be infused intravenously on Day 0. The first four patients enrolled will receive a single dose of 2 million cells/Kg and the last six patients enrolled, will receive a single dose of 5 million cells/kg.
  Interventions: Biological: Fucosylated MSC for Osteoporosis

INTERVENTIONS:
Biological: Fucosylated MSC for Osteoporosis — Aproximately 30 days before the infusion of the investigational product, patient bone marrow will be obtained according to standard practice of the Haematology University Hospital Virgen de la Arrixaca (HCUVA).
  Mononuclear bone marrow cells will be separated and cultured in GMP conditions to purify and obtain mesenchymal cell established dose range. The infusion day BM-MSCs will be fucosylated and resuspended in saline to a concentration of 5 million cells per 1 mL. Then, the final product will be packaged in syringes for intravenous administration to patients through a peripheral venous access.

SUMMARY:
The purpose of this study is to evaluate the safety of intravenous infusion of fucosylated autologous bone marrow cells as a new therapy in patients with established osteoporosis by a prospective, single-center, open, non-randomized and unblinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established osteoporosis according to standard clinical criteria.
* Patients who give their written informed consent to participate in the study consent.
* Meet all the inclusion criteria

Exclusion Criteria:

* Patients with concomitant systemic disease in the opinion of the investigator.
* Patients with rheumatoid arthritis, ankylosing spondylitis, chronic polyarticular arthritis.
* Current patients with neoplasm or history of any malignancy in the last 10 years except basal carcinoma or epidermoid skin.
* Patients with genetic disorders that are associated with secondary osteoporosis: Hemochromatosis, hypophosphatasia, osteogenesis imperfecta, Ehlers-Danlos syndrome, Marfan syndrome, Riley Day, porphyria, storage diseases syndrome.
* Patients receiving immunosuppressive chemotherapy or that could interfere with the process of cell proliferation.
* Transplant patients: bone marrow, kidney, liver, heart, lung.
* Patients with clinical criteria and anesthetics that contraindicate well sedation or bone marrow extraction.
* Patients participating in a clinical trial in the last 6 months.
* Patients with positive serology for hepatitis B, hepatitis C or HIV.
* Patients with inability to understand informed consent.
* Patients who are pregnant or breast-feeding actively.
* Patients physically fertile, defined as all women physiologically capable of becoming pregnant, UNLESS they are using reliable methods of contraception.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Rate of serious and non-serious adverse events related to the procedure. | 24 months from baseline
  During time frame the following items will be considered:
  Adverse effects related to the infusion moment. Occurrence of infectious complications after infusion of mesenchymal stem cells, because of the immunosuppressive effect of these cells.
  Appearance of procedure-related neoplasias.

SECONDARY OUTCOMES:
Number of new fractures | 24 months from baseline
Pain, measured by Visual Analog Scale | 24 months from baseline
  To measure pain, visual analogue scale (VAS) was used where 0 is no pain and 10 the worst pain imaginable.
Functionality, measured by Oswestry Disability Questionnaire | 24 months from baseline
  To identify the functional repercussion of lumbar pain, Oswestry Disability Questionnaire for back pain or Oswestry Disability Index is used.
Quality of Life, measured by EuroQoL-5D test | 24 months from baseline
  To measure the quality of life EuroQoL-5D psychometric test is used.
Bone resorption, measured by biochemical index | 24 months from baseline
  Aminoterminal telopeptide of type 1 collagen in the serum (serum NTX) (%) by ELISA technique.
Bone formation, measured by biochemical index | 24 months from baseline
  Osteocalcin in the serum by ELISA (BPG serum) (ng / mL) .
Bone formation, measured by biochemical index | 24 months from baseline
  Bone specific alkaline phosphatase in the serum by ELISA (serum FAO) (ug / L)
Bone formation, measured by biochemical index | 24 months from baseline
  Aminoterminal propeptide of procollagen type 1 in the serum by ELISA (serum P1NP) (ng / mL)
Bone metabolism, measured by biochemical index | 24 months from baseline
  Osteoprotegerin (OPG) (pmol / L) in the serum by ELISA.
Bone metabolism, measured by biochemical index | 24 months from baseline
  Ligand receptor activator of nuclear factor KB (RANKL) (pmol / L) in the serum by ELISA.
Bone Mineral Density , measured by dual energy x-ray absorptiometry (DXA) | 24 months from baseline
Bone structure, measured by histomorphometric evaluation | baseline and 4 months from baseline
Trabecular bone density measured by quantitative computed tomography of the radius | 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Linares Ferrando, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Virgen de la Arrixaca, El Palmar, Murcia, Spain